CLINICAL TRIAL: NCT06309628
Title: Analysis of Volatile Organic Compounds in the Breath of Lung Transplant Rejection
Brief Title: Analysis of Volatile Organic Compounds in the Breath of Lung Transplant Rejection Patients Using Infrared Spectroscopy
Status: Terminated | Type: Observational
Why Stopped: Interim determination of missed feasibility goals
Sponsor: Paragonix Technologies (Industry)
Collaborators: Breathe BioMedical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PGX-006
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Lung Transplant Rejection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A sample of the subject's breath, exhaled into a tube.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lung Transplant patients at risk for rejection: Patients who have had a lung transplant and are getting a bronchoscopy to test for rejection will provide a breathe sample. Once their rejection results come back after their sample has been collected their breathe samples will be sorted into rejection and non-rejection groups for analysis. All patients will have the same experiences in the study.
  Interventions: Diagnostic Test: Breathe sample

INTERVENTIONS:
Diagnostic Test: Breathe sample — Patients will provide two breathe sample into the Breathe device to see if their VOC patterns can be used to diagnose lung transplant rejection.

SUMMARY:
This study will sample and analyze volatile organic compounds (VOCs) from participants considered to be at risk for developing rejection following lung transplant by using infrared spectroscopy.

DETAILED DESCRIPTION:
The aim of this study is to sample and analyze volatile organic compounds (VOCs) from participants considered to be at risk for developing rejection following lung transplant. By using infrared spectroscopy, the breath sample analysis will help investigators describe and identify patterns of VOCs that are over- or under-represented in patients with post-lung transplant rejection when compared to the breath profiles of those without rejection. It is hypothesized that the profile of volatile chemicals in the breath of patients in the early stages of rejection will differ significantly from those individuals without rejection.

Primary objective

• To analyze the breath-born VOCs in breath profiles of lung transplant patients with rejection in comparison to lung transplant patients without rejection using infrared spectroscopy to determine the presence of lung rejection and to develop mathematical/statistical models of infrared absorption spectrum for identification of rejection.

Secondary objective

* To determine the best method to classify health status based on VOC data of breath samples
* To validate early test results on an additional infrared spectroscopic analyzer in post-lung transplant patients

The study is an unblinded, prospective case-control study. The study cohorts will include: 1) patients with confirmed post-lung transplant rejection via biopsy, and 2) control patients who have undergone lung transplant but are free from rejection as confirmed via biopsy. Breath samples collected from participants will be analyzed to characterize and further identify differences in infrared absorption profiles from each cohort using infrared spectroscopy. The data will be used to validate a previously developed machine learning algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patient is able to give informed consent
* Lung transplant patient who had both lungs transplanted
* Patient is at least 90 days after their lung transplant
* Patient is able to provide a breath sample

Exclusion Criteria:

* Patient is less than 18 years old
* Patient received multiple organ transplants
* Patient had an organ transplant prior to their lung transplant
* Patients who received a single lung transplant
* Patient less than 90 days or more than 1 year from their lung transplant
* If patient has smoked 4 hours or less before breath sample or consumed alcohol (including mouthwash) 8 hours or less before breath sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients who are receiving a bronchoscopy at least 90 days after a lung transplant.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Volatile Organic Compound profile | three to twelve months post-transplant
  The VOCs in the breath of patients experiencing lung rejection post-transplant per bronchoscopy will be compared to lung transplant patients who are not experiencing rejection

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hartwig, MD, Principal Investigator — Duke University; Matthew Pipeling, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States